CLINICAL TRIAL: NCT00439478
Title: The Dental Safety Profile of High-Dose Radioiodine Therapy for Thyroid Cancer
Brief Title: Dental Safety Profile of High-Dose Radioiodine Therapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 171074
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-10

CONDITIONS: Thyroid Cancer
Keywords: Radioiodine, Thyroid Cancer, Sialadenitis, Xerostomia
MeSH Terms: conditions — Thyroid Neoplasms; Sialadenitis; Xerostomia | interventions — Iodine-131

INTERVENTIONS:
Drug: Radioiodine

SUMMARY:
We aim to assess the incidence of oral and dental adverse events after high-dose radioiodine therapy for differentiated thyroid cancer.

DETAILED DESCRIPTION:
Sialadenitis and xerostomia are the most frequent adverse events of high-dose radioiodine therapy. Saliva has vital functions in maintaining periodontal and oral health. Therefore, xerostomia not only impairs quality of life permanently, but may also increase the risk of caries and tooth extractions. Nevertheless, despite more than 6 decades of radioiodine therapy for thyroid cancer, large studies on long-term oral adverse events are still lacking. In the present study, we investigate the influence of high-dose radioiodine therapy on the long-term oral health.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed differentiated thyroid cancer
* status after total thyroidectomy
* status after subsequent high-dose radioiodine treatment
* regular follow-up by a board-certified dentist
* a minimum follow-up of 1 year after radioiodine therapy.

Exclusion Criteria:

* anaplastic thyroid cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202
Dates: Start 2004-09; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beat Müller, MD, Study Director — Division of Endocrinology, University Hospital Basel
Locations (1):
- University Hospital, Basel, Switzerland